CLINICAL TRIAL: NCT01397565
Title: Minilaparoscopic Versus Conventional Laparoscopic Cholecystectomy: A Randomized Trial
Brief Title: Minilaparoscopic Versus Conventional Laparoscopic Cholecystectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Dr. Liane S. Feldman, MD, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11-053-SDR
Record Dates: First submitted 2011-07-05; First posted 2011-07-19 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Cholelithiasis; Cholecystectomy
Keywords: Cholecystectomy; Laparoscopy; Minilaparoscopic surgery; Post-operative pain; Recovery time
MeSH Terms: conditions — Cholelithiasis; Pain, Postoperative | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laparoscopic cholecystectomy (Active Comparator): Patients in this arm will undergo conventional laparoscopic cholecystectomy
  Interventions: Procedure: Laparoscopic cholecystectomy
- Minilaparoscopic cholecystectomy (Experimental): Patients in this arm will undergo laparoscopic cholecystectomy using minilaparoscopic instruments
  Interventions: Procedure: Minilaparoscopic cholecystectomy

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy — Laparoscopic cholecystectomy
  Arms: Laparoscopic cholecystectomy
Procedure: Minilaparoscopic cholecystectomy — Laparoscopic cholecystectomy performed using minilaparoscopic instruments
  Other Names: Needlescopic surgery
  Arms: Minilaparoscopic cholecystectomy

SUMMARY:
Laparoscopic cholecystectomy is one of the most commonly performed operations in general surgery and is considered the standard of care for cholecystectomy for benign biliary disease. The laparoscopic approach to cholecystectomy, when compared to open surgery, is associated with less postoperative pain, quicker recovery time and an improved cosmetic result.

Most commonly, laparoscopic cholecystectomy is performed using a 10-12mm port in the umbilicus with 3 additional ports consisting of either three 5mm ports, or a combination of two 5mm ports and one 10mm port. A new technique called minilaparoscopic (also referred to as needlescopic) surgery has recently emerged. Minilaparoscopic surgery replaces 5mm trocars with smaller 3mm trocars. Surgery using these smaller trocars is hypothesized to further reduce postoperative pain and recovery time as well as improve cosmetic results following laparoscopic surgery. Our goal is to compare these outcomes in a randomized trial comparing conventional to minilaparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Background Since its introduction in the late 1980's, laparoscopic cholecystectomy has quickly become the standard of care in surgery for benign disease of the gallbladder. When compared to open surgery, laparoscopic surgery is associated with decreased post-operative pain. Recovery time and return to usual activity are also significantly shorter following the laparoscopic procedure. Cholecystectomy in the era of laparoscopic surgery has become an out-patient procedure. Furthermore, laparoscopic surgery eliminates a large surgical scar and provides patients an improved cosmetic result .

Laparoscopic technology has evolved rapidly over the last 20 years. The quality of instruments, and especially of optics, has greatly improved since the first laparoscopic cholecystectomies were performed. A significant trend in the development of new technologies has been the move toward smaller instruments and cameras. Where 10mm cameras were standard in the early years of laparoscopy, 5mm cameras now offer excellent optical quality and permit the use of fewer 10mm trocars. In this movement toward increasingly less invasive techniques, minilaparoscopic surgery has emerged. Minilaparoscopic surgery (also called needlescopic surgery) involves the use of smaller trocars and instruments, typically 3mm in size. It is hypothesized that smaller trocars cause less tissue damage and therefore result in improved post-operative pain and recovery, while offering the additional benefit of improved cosmesis.

Previous studies have found minilaparoscopic surgery to be safe, with complication rates no greater than those of conventional laparoscopic technique. In some studies, minilaparoscopic cholecystectomy has been associated with slightly increased operative time. Previous studies have also noted higher conversion rates (a change in the planned operative technique to another technique), however this conversion is typically from minilaparoscopy to conventional laparoscopy; the rate of conversion from minilaparoscopy to an open procedure is no higher than with conventional laparoscopy. However a recent meta-analysis performed by Thakur et al. (1) found that while some studies have shown these trends toward longer operative times and increased conversion rates, the overall evidence for this is weak.

While a number of previous studies have attempted evaluate the benefits that patients derive from minilaparoscopic surgery, including post-operative pain and recovery time, many of these studies have been flawed by methodological concerns. Thakur et al showed in their meta-analysis that minilaparoscopic cholecystectomy was associated with improved cosmesis at one month as well as reduced post-operative pain and faster recovery time. These benefits however were estimated to be minimal based on the available evidence. Unclear reporting of trials and flawed study design, specifically the lack of "intention to treat" analysis, make the interpretation of available data difficult and the meta-analysis concluded that "the evidence for using minicholecystecomy is unclear."

More high quality evidence is needed for the surgical community to determine the utility and benefits of minilaparoscopic cholecystectomy. It is our hope that through a rigorous methodological design we can add to the available literature and determine if minilaparoscopic cholecystectomy is a valuable technique that will benefit patients.

Hypothesis Minilaparoscopic surgery will reduce postoperative pain and recovery time, as well as improve cosmetic results in patients undergoing cholecystectomy.

Objectives

A randomized trial comparing minilaparoscopic cholecystectomy to standard laparoscopic cholecystectomy will be performed to:

1. Determine if minilaparoscopic surgery is associated with decreased postoperative pain
2. Determine if minilaparoscopic surgery results is associated with quicker recovery and return to usual activities
3. Determine if minilaparoscopic surgery is associated with in an improved cosmetic result

ELIGIBILITY:
Inclusion Criteria:

* minimum 18 years of age
* referred for elective cholecystectomy for benign biliary stone disease

Exclusion Criteria:

* previous upper gastrointestinal surgery
* acute cholecystitis (past or present)
* American Society of Anesthesiologists (ASA) class greater than or equal to 4
* pregnancy
* morbid obesity (BMI > 35 kg/m2)
* inability to comprehend questionnaires in either English or French
* psychiatric conditions that preclude cooperation and/or comprehension of questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2012-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Post-operative pain | First seven days post-op, 3 weeks post-op
  Post-operative pain will be assessed during the first week post-operatively using a diary that will be provided to patients. In this diary, patients will score their pain daily using a visual analog scale (0=no pain and 10=severe pain) and record use of pain medications for the first seven days post-operatively. Patients will again be asked to score their pain using the visual analog scale at the regularly scheduled follow-up visit three weeks post-op.
Time to recovery | 3 weeks post-operatively
  Time to recovery (return to baseline level of activity) will be evaluated by comparing baseline physical activity scores to physical activity scores determined at the follow-up visit three weeks post-op. Physical activity scores will be obtained using the validated CHAMPS questionnaire (2)
Cosmetic result | 3 months post-operatively
  Cosmetic result will be evaluated using a scar assessment questionnaire (3), that will be administered by the study coordinator at the routine post-op visit as well as at three months by telephone

SECONDARY OUTCOMES:
Operative complications | First 3 months post-op
  Intra-operative, in-hospital (if applicable) and postoperative complications will be recorded and graded according to the Clavien Classification. Superficial and deep incisional surgical site infections will be defined according to the CDC definition.
Operative technique | Recorded at visit 3 weeks post-op
  Conversion to conventional laparoscopic technique or open procedure will be recorded at the time of operation.
Length of operation | Recorded at visit 3 weeks post-op
  The time necessary to complete the intervention will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Liane Feldman, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Background] Thakur V, Schlachta CM, Jayaraman S. Minilaparoscopic versus conventional laparoscopic cholecystectomy a systematic review and meta-analysis. Ann Surg. 2011 Feb;253(2):244-58. doi: 10.1097/SLA.0b013e318207bf52. PMID 21183848
- [Background] Feldman LS, Kaneva P, Demyttenaere S, Carli F, Fried GM, Mayo NE. Validation of a physical activity questionnaire (CHAMPS) as an indicator of postoperative recovery after laparoscopic cholecystectomy. Surgery. 2009 Jul;146(1):31-9. doi: 10.1016/j.surg.2009.02.019. PMID 19541008
- [Background] Durani P, McGrouther DA, Ferguson MW. The Patient Scar Assessment Questionnaire: a reliable and valid patient-reported outcomes measure for linear scars. Plast Reconstr Surg. 2009 May;123(5):1481-1489. doi: 10.1097/PRS.0b013e3181a205de. PMID 19407619
- [Derived] Alhashemi M, Almahroos M, Fiore JF Jr, Kaneva P, Gutierrez JM, Neville A, Vassiliou MC, Fried GM, Feldman LS. Impact of miniport laparoscopic cholecystectomy versus standard port laparoscopic cholecystectomy on recovery of physical activity: a randomized trial. Surg Endosc. 2017 May;31(5):2299-2309. doi: 10.1007/s00464-016-5232-z. Epub 2016 Sep 21. PMID 27655375